CLINICAL TRIAL: NCT07214805
Title: Understanding Perceptions of and Reactions to Ultra-processed Food Label Designs
Brief Title: Perceptions of and Reactions to Ultra-Processed Menu Label Designs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00034378-2; 5R01DK139327-02 (NIH)
Record Dates: First submitted 2025-10-06; First posted 2025-10-09 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Food Choices
Keywords: food labeling; ultra-processed foods
MeSH Terms: interventions — Dyrk Kinases

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to view a fast-food online ordering menu with one of sixteen labeling schemes, varying by message ("Ultra-Processed" vs. "Contains Food Additives" vs. "Warning: Ultra-Processed" vs. "Warning: UPF"), background and text color (red with white text vs. yellow with black text), and type (icon-plus-text vs. text-only). Participants will be asked about a hypothetical intention to purchase a menu item with the label to which the participants were randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (16):
- Ultra-Processed, Red, Icon-plus-text Labels (Experimental): A red icon-plus-text label that reads "ULTRA-PROCESSED" in white text will be placed beneath ultra-processed menu items. Labels will include a triangle icon with an exclamation point directly preceding the label text.
  Interventions: Behavioral: Ultra-Processed, Red, Icon-plus-text Labels
- Contains Food Additives, Red, Icon-plus-text Labels (Experimental): A red icon-plus-text label that reads "CONTAINS FOOD ADDITIVES" in white text will be placed beneath ultra-processed menu items. Labels will include a triangle icon with an exclamation point directly preceding the label text.
  Interventions: Behavioral: Contains Food Additives, Red, Icon-plus-text Labels
- Warning Ultra-Processed, Red, Icon-plus-text Labels (Experimental): A red icon-plus-text label that reads "WARNING: ULTRA-PROCESSED" in white text will be placed beneath ultra-processed menu items. Labels will include a triangle icon with an exclamation point directly preceding the label text.
  Interventions: Behavioral: Warning Ultra-Processed, Red, Icon-plus-text Labels
- Warning UPF, Red, Icon-plus-text Labels (Experimental): A red icon-plus-text label that reads "WARNING: UPF" in white text will be placed beneath ultra-processed menu items. Labels will include a triangle icon with an exclamation point directly preceding the label text.
  Interventions: Behavioral: Warning UPF, Red, Icon-plus-text Labels
- Ultra-Processed, Yellow, Icon-plus-text Labels (Experimental): A yellow icon-plus-text label that reads "ULTRA-PROCESSED" in black text will be placed beneath ultra-processed menu items. Labels will include a triangle icon with an exclamation point directly preceding the label text.
  Interventions: Behavioral: Ultra-Processed, Yellow, Icon-plus-text Labels
- Contains Food Additives, Yellow, Icon-plus-text Labels (Experimental): A yellow icon-plus-text label that reads "CONTAINS FOOD ADDITIVES" in black text will be placed beneath ultra-processed menu items. Labels will include a triangle icon with an exclamation point directly preceding the label text.
  Interventions: Behavioral: Contains Food Additives, Yellow, Icon-plus-text Labels
- Warning Ultra-Processed, Yellow, Icon-plus-text Labels (Experimental): A yellow icon-plus-text label that reads "WARNING: ULTRA-PROCESSED" in black text will be placed beneath ultra-processed menu items. Labels will include a triangle icon with an exclamation point directly preceding the label text.
  Interventions: Behavioral: Warning Ultra-Processed, Yellow, Icon-plus-text Labels
- Warning UPF, Yellow, Icon-plus-text Labels (Experimental): A yellow icon-plus-text label that reads "WARNING: UPF" in black text will be placed beneath ultra-processed menu items. Labels will include a triangle icon with an exclamation point directly preceding the label text.
  Interventions: Behavioral: Warning UPF, Yellow, Icon-plus-text Labels
- Ultra-Processed, Red, Text-only Labels (Experimental): A red text-only label that reads "ULTRA-PROCESSED" in white text will be placed beneath ultra-processed menu items.
  Interventions: Behavioral: Ultra-Processed, Red, Text-only Labels
- Contains Food Additives, Red, Text-only Labels (Experimental): A red text-only label that reads "CONTAINS FOOD ADDITIVES" in white text will be placed beneath ultra-processed menu items.
  Interventions: Behavioral: Contains Food Additives, Red, Text-only Labels
- Warning Ultra-Processed, Red, Text-only Labels (Experimental): A red text-only label that reads "WARNING: ULTRA-PROCESSED" in white text will be placed beneath ultra-processed menu items.
  Interventions: Behavioral: Warning Ultra-Processed, Red, Text-only Labels
- Warning UPF, Red, Text-only Labels (Experimental): A red text-only label that reads "WARNING: UPF" in white text will be placed beneath ultra-processed menu items.
  Interventions: Behavioral: Warning UPF, Red, Text-only Labels
- Ultra-Processed, Yellow, Text-only Labels (Experimental): A yellow text-only label that reads "ULTRA-PROCESSED" in black text will be placed beneath ultra-processed menu items.
  Interventions: Behavioral: Ultra-Processed, Yellow, Text-only Labels
- Contains Food Additives, Yellow, Text-only Labels (Experimental): A yellow text-only label that reads "CONTAINS FOOD ADDITIVES" in black text will be placed beneath ultra-processed menu items.
  Interventions: Behavioral: Contains Food Additives, Yellow, Text-only Labels
- Warning Ultra-Processed, Yellow, Text-only Labels (Experimental): A red text-only label that reads "WARNING: ULTRA-PROCESSED" in black text will be placed beneath ultra-processed menu items.
  Interventions: Behavioral: Warning Ultra-Processed, Yellow, Text-only Labels
- Warning UPF, Yellow, Text-only Labels (Experimental): A yellow text-only label that reads "WARNING: UPF" in black text will be placed beneath ultra-processed menu items.
  Interventions: Behavioral: Warning UPF, Yellow, Text-only Labels

INTERVENTIONS:
Behavioral: Ultra-Processed, Red, Icon-plus-text Labels — Participants will view a fast-food restaurant menu excerpt. Each menu item will be displayed with an image of the item, name, price, and total calories. The Ultra-Processed, Red, Icon-plus-text labels will be displayed next to items that are ultra-processed. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Ultra-Processed, Red, Icon-plus-text Labels
Behavioral: Contains Food Additives, Red, Icon-plus-text Labels — Participants will view a fast-food restaurant menu excerpt. Each menu item will be displayed with an image of the item, name, price, and total calories. The Contains Food Additives, Red, Icon-plus-text labels will be displayed next to items that are ultra-processed. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Contains Food Additives, Red, Icon-plus-text Labels
Behavioral: Warning Ultra-Processed, Red, Icon-plus-text Labels — Participants will view a fast-food restaurant menu excerpt. Each menu item will be displayed with an image of the item, name, price, and total calories. The Warning Ultra-Processed, Red, Icon-plus-text labels will be displayed next to items that are ultra-processed. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Warning Ultra-Processed, Red, Icon-plus-text Labels
Behavioral: Warning UPF, Red, Icon-plus-text Labels — Participants will view a fast-food restaurant menu excerpt. Each menu item will be displayed with an image of the item, name, price, and total calories. The Warning UPF, Red, Icon-plus-text labels will be displayed next to items that are ultra-processed. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Warning UPF, Red, Icon-plus-text Labels
Behavioral: Ultra-Processed, Yellow, Icon-plus-text Labels — Participants will view a fast-food restaurant menu excerpt. Each menu item will be displayed with an image of the item, name, price, and total calories. The Ultra-Processed, Yellow, Icon-plus-text labels will be displayed next to items that are ultra-processed. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Ultra-Processed, Yellow, Icon-plus-text Labels
Behavioral: Contains Food Additives, Yellow, Icon-plus-text Labels — Participants will view a fast-food restaurant menu excerpt. Each menu item will be displayed with an image of the item, name, price, and total calories. The Contains Food Additives, Yellow, Icon-plus-text labels will be displayed next to items that are ultra-processed. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Contains Food Additives, Yellow, Icon-plus-text Labels
Behavioral: Warning Ultra-Processed, Yellow, Icon-plus-text Labels — Participants will view a fast-food restaurant menu excerpt. Each menu item will be displayed with an image of the item, name, price, and total calories. The Warning Ultra-Processed, Yellow, Icon-plus-text labels will be displayed next to items that are ultra-processed. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Warning Ultra-Processed, Yellow, Icon-plus-text Labels
Behavioral: Warning UPF, Yellow, Icon-plus-text Labels — Participants will view a fast-food restaurant menu excerpt. Each menu item will be displayed with an image of the item, name, price, and total calories. The Warning UPF, Yellow, Icon-plus-text labels will be displayed next to items that are ultra-processed. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Warning UPF, Yellow, Icon-plus-text Labels
Behavioral: Ultra-Processed, Red, Text-only Labels — Participants will view a fast-food restaurant menu excerpt. Each menu item will be displayed with an image of the item, name, price, and total calories. The Ultra-Processed, Red, Text-only labels will be displayed next to items that are ultra-processed. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Ultra-Processed, Red, Text-only Labels
Behavioral: Contains Food Additives, Red, Text-only Labels — Participants will view a fast-food restaurant menu excerpt. Each menu item will be displayed with an image of the item, name, price, and total calories. The Contains Food Additives, Red, Text-only labels will be displayed next to items that are ultra-processed. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Contains Food Additives, Red, Text-only Labels
Behavioral: Warning Ultra-Processed, Red, Text-only Labels — Participants will view a fast-food restaurant menu excerpt. Each menu item will be displayed with an image of the item, name, price, and total calories. The Warning Ultra-Processed, Red, Text-only labels will be displayed next to items that are ultra-processed. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Warning Ultra-Processed, Red, Text-only Labels
Behavioral: Warning UPF, Red, Text-only Labels — Participants will view a fast-food restaurant menu excerpt. Each menu item will be displayed with an image of the item, name, price, and total calories. The Warning UPF, Red, Text-only labels will be displayed next to items that are ultra-processed. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Warning UPF, Red, Text-only Labels
Behavioral: Ultra-Processed, Yellow, Text-only Labels — Participants will view a fast-food restaurant menu excerpt. Each menu item will be displayed with an image of the item, name, price, and total calories. The Ultra-Processed, Yellow, Text-only labels will be displayed next to items that are ultra-processed. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Ultra-Processed, Yellow, Text-only Labels
Behavioral: Contains Food Additives, Yellow, Text-only Labels — Participants will view a fast-food restaurant menu excerpt. Each menu item will be displayed with an image of the item, name, price, and total calories. The Contains Food Additives, Yellow, Text-only labels will be displayed next to items that are ultra-processed. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Contains Food Additives, Yellow, Text-only Labels
Behavioral: Warning Ultra-Processed, Yellow, Text-only Labels — Participants will view a fast-food restaurant menu excerpt. Each menu item will be displayed with an image of the item, name, price, and total calories. The Warning Ultra-Processed, Yellow, Text-only labels will be displayed next to items that are ultra-processed. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Warning Ultra-Processed, Yellow, Text-only Labels
Behavioral: Warning UPF, Yellow, Text-only Labels — Participants will view a fast-food restaurant menu excerpt. Each menu item will be displayed with an image of the item, name, price, and total calories. The Warning UPF, Yellow, Text-only labels will be displayed next to items that are ultra-processed. Participants will view the menu and then the label in isolation and then be asked about a hypothetical intention to purchase a menu item with the label.
  Arms: Warning UPF, Yellow, Text-only Labels

SUMMARY:
The primary objective of this study is to explore perceptions and understanding of different menu label designs related to ultra-processed foods (UPF). Participants will be randomized to view a fast-food online menu excerpt featuring one of sixteen labeling conditions and then will answer questions about the participant's reactions to and interpretations of the label, perceived label effectiveness, the intention to purchase a menu item with the label, as well as the participant's perceptions of fast-food menu items with and without the label.

DETAILED DESCRIPTION:
This survey will explore the perceptions and understanding of different hypothetical UPF menu label designs. The survey research firm CloudResearch will recruit a sample of ~12,400 adults aged 18 years and older who reside in the United States.

This exploratory study will use a factorial experiment to assess different UPF label designs. Participants will be randomized to view a fast-food menu excerpt with one of sixteen labeling schemes, varying by message ("Ultra-Processed" vs. "Contains Food Additives" vs. "Warning: Ultra-Processed" vs. "Warning: UPF"), background and text color (red background with white text vs. yellow background with black text), and type (icon-plus-text vs. text-only). All menus will consist of a selection of food and beverage items, and select items will have the UPF label.

Participants will be shown the menu and the label in isolation and will then be asked about the participant's interpretations of the label, reactions to the label, perceived message effectiveness (PME) of the label, how helpful the participant finds the label to be, and the participant's intention to purchase a menu item with the label. The participants will also be shown two different individual fast-food items with the label to which the participant was randomized in random order and asked about the perceived appeal and healthfulness of the menu items.

The primary outcome will be intention to purchase a hypothetical menu item with the label. Secondary outcomes include label interpretation, perceived label understandability, perceived label believability, perception that the label grabbed attention, perceived message effectiveness (PME) of the label, perceived helpfulness of the label. Other outcomes include perceived level of appeal of menu items, and perceived level of healthfulness of menu items.

ELIGIBILITY:
Inclusion Criteria:

* - 18 years of age or older
* Member of the CloudResearch panel
* Residing in the United States

Exclusion Criteria:

* <18 years of age
* Not residing in the United States
* Completed the survey implausibly quickly based on the distribution of the time to complete the survey among all participants
* Failed the built-in Qualtrics survey fraud detection measures
* Failed attention check question included in the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14720 (Actual)
Dates: Start 2025-10-09 (Actual); Primary Completion 2025-11-02 (Actual); Study Completion 2025-11-02 (Actual)

PRIMARY OUTCOMES:
Intention to purchase | Immediately after viewing the menu excerpt and label image
  Intention to purchase is measured with the survey question: "How likely would you be to purchase a menu item with this label?" Response options are a 5-point Likert scale: 1=Very unlikely, 2=Unlikely, 3=Somewhat unlikely, 4=Neither likely nor unlikely, 5=Somewhat likely, 6=Likely, 7=Very likely. A higher rating is better.

SECONDARY OUTCOMES:
Label interpretation | Immediately after viewing the menu excerpt and label
  Label interpretation is assessed with the survey question: "Imagine that you are in a fast-food restaurant (such as Dunkin') to order for yourself. Next, is a question about the label, as displayed on the menu example. If you saw this label next to an item on the menu, what would you think the label indicates about the item? [check all that apply]". Response options provided are a range of statements about the menu item, including 1="This menu item is unhealthy", 2="This menu item contains artificial ingredients", 3="This menu item used a lot of natural resources to produce", 4="This menu item will keep you full for a long time", 5="This menu item is bad for the environment, 6="This menu item costs more", 7="This menu item was made using industrial processing techniques", "This menu item is high in (8) sugar (9) sodium, (10) saturated fat, (11) calories". Also included are "I don't know" and an "Other" option with open-text entry.
Perceived label understandability | Immediately after viewing the menu excerpt and label image
  After viewing the label, participants will be asked how much the participant agrees or disagrees with the following statement: "This label is easy to understand". Response options are a unipolar 5-point Likert scale: 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=A great deal. A higher ranking is better.
Perceived label believability | Immediately after viewing the menu excerpt and label image
  After viewing the label, participants will be asked how much the participant agrees or disagrees with the following statement: "This label is believable to me". Response options are a unipolar 5-point Likert scale: 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=A great deal. A higher ranking is better.
Perception that label grabbed attention | Immediately after viewing the menu excerpt and label image
  After viewing the label, participants will be asked how much the participant agrees or disagrees with the following statement: "This label grabs my attention". Response options are a unipolar 5-point Likert scale: 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=A great deal. A higher ranking is better.
Perceived message effectiveness (PME) as assessed by the University of North Carolina (UNC)-PME scale | Immediately after viewing the menu excerpt and label image
  Perceived message effectiveness (PME) is measured using the unipolar 3-item University of North Carolina (UNC)-PME scale. Participants will be asked how much each label discourages consumption of or evokes concern of unpleasantness about consumption of foods with the label. After viewing the label, participants will be asked how much the participant agrees or disagrees with the following statements: "This label discourages me from wanting to eat foods with this label", "This label makes foods with this label seem unpleasant", and "This label makes me concerned about the health effects of eating menu items with this label". Response options are a 5-point Likert scale: 1=Not at all, 2=A little bit, 3=Somewhat, 4=Quite a bit, 5=A great deal. A higher ranking is better.
Perceived label helpfulness | Immediately after viewing the menu excerpt and label image
  Perceived label helpfulness is measured with the survey question: "How helpful would you find this label when deciding what to order at a fast-food restaurant?" Response options are a 7-point Likert scale: 1=Very unhelpful, 2=Unhelpful, 3=Somewhat unhelpful, 4=Neither helpful nor unhelpful, 5=Somewhat helpful, 6=Helpful, 7=Very helpful. A higher ranking is better.

OTHER OUTCOMES:
Perceived level of appeal of labeled food item | Immediately after viewing each menu item
  Perceived level of appeal of food item is measured after showing participants two different individual menu items separately by label condition. After showing each item, the survey question asks, "How appealing do you think this item is?", and response options are a 7-point Likert scale: 1=Very unappealing, 2=Unappealing, 3=Slightly unappealing, 4=Neither appealing nor unappealing, 5=Slightly appealing, 6=Appealing, 7=Very appealing. A higher ranking is better
Perceived level of healthfulness of labeled food item | Immediately after viewing each menu item
  Perceived level of healthfulness of labeled food item is measured after showing participants two different individual menu items separately by label condition. After showing each item, the survey question asks, "How healthy do you think this item is?", and response options are a 7-point Likert scale: 1=Very unhealthy, 2=Unhealthy, 3=Slightly unhealthy, 4=Neither unhealthy nor healthy, 5=Slightly healthy, 6=Healthy, 7=Very healthy. A higher ranking is better.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Wolfson, PhD, MPP, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share anonymous individual level data with members of the research team and with other interested researchers upon request. After results have been published the investigators will make study data available on Open Science Framework consistent with the Data Sharing and Management Plan.
Supporting Information: SAP, Analytic Code
Time Frame: After the study team has published results, data and other documents will be made available. There is no end date for availability.
Access Criteria: Data and supporting documentation will be publicly available on the Open Science Framework website.